CLINICAL TRIAL: NCT00737100
Title: A Randomized, Double-blind, Placebo-controlled Parallel Group Study to Investigate the Safety and Efficacy of Two Doses of Tiotropium Bromide (2.5 mcg and 5 mcg) Administered Once Daily Via the Respimat Device for 12 Weeks in Patients With Cystic Fibrosis.
Brief Title: Safety and Efficacy of 12-wk Treatment With Two Doses of Tiotropium Respimat in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.339; 2008-001156-43 (EudraCT Number: EudraCT)
Expanded Access: Available
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Results first posted 2011-04-13 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tiotropium Bromide

ARMS (3):
- Tiotropium Respimat 2.5 mcg (Experimental): patient to receive low dose tiotropium once daily
  Interventions: Drug: tiotropium bromide-low dose-2.5mcg
- Tiotropium Respimat 5 mcg (Experimental): patient to receive high dose tiotropium once daily
  Interventions: Drug: Tiotropium bromide 5 mcg
- Placebo Respimat (Placebo Comparator): patient to receive placebo once daily
  Interventions: Drug: Placebo Respimat

INTERVENTIONS:
Drug: Placebo Respimat — patient to receive placebo matching active drug once daily
  Arms: Placebo Respimat
Drug: Tiotropium bromide 5 mcg — patient to recieve high dose tiotropium once daily
  Arms: Tiotropium Respimat 5 mcg
Drug: tiotropium bromide-low dose-2.5mcg — patient to receive low dose tiotropium once daily
  Arms: Tiotropium Respimat 2.5 mcg

SUMMARY:
This study evaluates the effects of 12-week treatment with two doses of tiotropium bromide (2.5 mcg q.d. and 5 mcg q.d.) compared to placebo administered via the Respimat device on lung function in patients with Cystic Fibrosis. The selection of the optimal dose will be based on bronchodilator efficacy, safety evaluations and pharmacokinetic evaluations

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients
2. Diagnosis of Cystic Fibrosis (positive sweat chloride test or two identifiable mutations)
3. Pre-bronchodilator FEV1 greater/equal 25% of predicted values

Exclusion criteria:

1. Significant history of allergy/hypersensitivity
2. Hypersensitivity to study drug
3. Participation in another trial
4. Female patients who are pregnant or lactating
5. Female patients of childbearing potential
6. Patients who have started a new medication for CF within 4 weeks of screening
7. Patients with known substance abuse
8. Clinically significant disease other than CF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (107):
- United States (26):
  - 205.339.006 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 205.339.019 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.339.023 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 205.339.021 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 205.339.030 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 205.339.031 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 205.339.014 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 205.339.022 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 205.339.013 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 205.339.001 Boehringer Ingelheim Investigational Site, Iowa City, Iowa
  - 205.339.017 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 205.339.025 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 205.339.016 Boehringer Ingelheim Investigational Site, Grand Rapids, Michigan
  - 205.339.018 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 205.339.029 Boehringer Ingelheim Investigational Site, Long Branch, New Jersey
  - 205.339.009 Boehringer Ingelheim Investigational Site, Morristown, New Jersey
  - 205.339.002 Boehringer Ingelheim Investigational Site, Syracuse, New York
  - 205.339.024 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 205.339.020 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.339.032 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.339.010 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.339.004 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 205.339.005 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 205.339.026 Boehringer Ingelheim Investigational Site, Colchester, Vermont
  - 205.339.011 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 205.339.003 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Australia (4):
  - 205.339.100 Boehringer Ingelheim Investigational Site, Westmead, New South Wales
  - 205.339.101 Boehringer Ingelheim Investigational Site, Westmead, New South Wales
  - 205.339.103 Boehringer Ingelheim Investigational Site, Adelaide, South Australia
  - 205.339.104 Boehringer Ingelheim Investigational Site, Subiaco, Western Australia
- Belgium (3):
  - 205.339.111 Boehringer Ingelheim Investigational Site, Brussels
  - 205.339.112 Boehringer Ingelheim Investigational Site, Jette
  - 205.339.110 Boehringer Ingelheim Investigational Site, Leuven
- France (32):
  - 205.339.3310A Boehringer Ingelheim Investigational Site, Amiens
  - 205.339.3317A Boehringer Ingelheim Investigational Site, Angers
  - 205.339.3317C Boehringer Ingelheim Investigational Site, Angers
  - 205.339.3317D Boehringer Ingelheim Investigational Site, Angers
  - 205.339.3317E Boehringer Ingelheim Investigational Site, Angers
  - 205.339.3314A Boehringer Ingelheim Investigational Site, Bron
  - 205.339.3314B Boehringer Ingelheim Investigational Site, Bron
  - 205.339.3314C Boehringer Ingelheim Investigational Site, Bron
  - 205.339.3302A Boehringer Ingelheim Investigational Site, Lille
  - 205.339.3302B Boehringer Ingelheim Investigational Site, Lille
  - 205.339.3302C Boehringer Ingelheim Investigational Site, Lille
  - 205.339.3303A Boehringer Ingelheim Investigational Site, Lisieux
  - 205.339.3304A Boehringer Ingelheim Investigational Site, Montpellier
  - 205.339.3304B Boehringer Ingelheim Investigational Site, Montpellier
  - 205.339.3308A Boehringer Ingelheim Investigational Site, Nantes
  - 205.339.3308B Boehringer Ingelheim Investigational Site, Nantes
  - 205.339.3308C Boehringer Ingelheim Investigational Site, Nantes
  - 205.339.3301B Boehringer Ingelheim Investigational Site, Paris
  - 205.339.3312A Boehringer Ingelheim Investigational Site, Paris
  - 205.339.3312C Boehringer Ingelheim Investigational Site, Paris
  - 205.339.3313A Boehringer Ingelheim Investigational Site, Paris
  - 205.339.3313B Boehringer Ingelheim Investigational Site, Paris
  - 205.339.3318A Boehringer Ingelheim Investigational Site, Rennes
  - 205.339.3318C Boehringer Ingelheim Investigational Site, Rennes
  - 205.339.3318G Boehringer Ingelheim Investigational Site, Rennes
  - 205.339.3315C Boehringer Ingelheim Investigational Site, Roscoff
  - 205.339.3315D Boehringer Ingelheim Investigational Site, Roscoff
  - 205.339.3306A Boehringer Ingelheim Investigational Site, Rouen
  - 205.339.3306B Boehringer Ingelheim Investigational Site, Rouen
  - 205.339.3307A Boehringer Ingelheim Investigational Site, Rouen
  - 205.339.3309A Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
  - 205.339.3316A Boehringer Ingelheim Investigational Site, Vannes
- Germany (11):
  - 205.339.49132 Boehringer Ingelheim Investigational Site, Erlangen
  - 205.339.49137 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.339.49133 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 205.339.49134 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 205.339.49131 Boehringer Ingelheim Investigational Site, Gerlingen
  - 205.339.49145 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.339.49135 Boehringer Ingelheim Investigational Site, Hanover
  - 205.339.49141 Boehringer Ingelheim Investigational Site, Heidelberg
  - 205.339.49140 Boehringer Ingelheim Investigational Site, München
  - 205.339.49142 Boehringer Ingelheim Investigational Site, München
  - 205.339.49130 Boehringer Ingelheim Investigational Site, Tübingen
- Italy (3):
  - 205.339.233 Boehringer Ingelheim Investigational Site, Ancona
  - 205.339.231 Boehringer Ingelheim Investigational Site, Florence
  - 205.339.234 Boehringer Ingelheim Investigational Site, Genova
- Netherlands (2):
  - 205.339.171 Boehringer Ingelheim Investigational Site, Groesbeek
  - 205.339.170 Boehringer Ingelheim Investigational Site, Rotterdam
- New Zealand (2):
  - 205.339.105 Boehringer Ingelheim Investigational Site, Grafton / Auckland
  - 205.339.106 Boehringer Ingelheim Investigational Site, Hamilton
- Portugal (4):
  - 205.339.221 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.339.225 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.339.223 Boehringer Ingelheim Investigational Site, Porto
  - 205.339.224 Boehringer Ingelheim Investigational Site, Porto
- Russia (8):
  - 205.339.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 205.339.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 205.339.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 205.339.07007 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 205.339.07005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.339.07006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.339.07008 Boehringer Ingelheim Investigational Site, Voronezh
  - 205.339.07004 Boehringer Ingelheim Investigational Site, Yaroslavl
- United Kingdom (12):
  - 205.339.44180 Boehringer Ingelheim Investigational Site, Belfast
  - 205.339.44190 Boehringer Ingelheim Investigational Site, Birmingham
  - 205.339.44193 Boehringer Ingelheim Investigational Site, Boston
  - 205.339.44192 Boehringer Ingelheim Investigational Site, Leeds
  - 205.339.44191 Boehringer Ingelheim Investigational Site, Lincoln
  - 205.339.44185 Boehringer Ingelheim Investigational Site, Liverpool
  - 205.339.44186 Boehringer Ingelheim Investigational Site, Liverpool
  - 205.339.44183 Boehringer Ingelheim Investigational Site, Nottingham
  - 205.339.44182 Boehringer Ingelheim Investigational Site, Oxford
  - 205.339.44194 Boehringer Ingelheim Investigational Site, Plymouth
  - 205.339.44181 Boehringer Ingelheim Investigational Site, Sheffield
  - 205.339.44184 Boehringer Ingelheim Investigational Site, Wolverhampton

REFERENCES:
- [Derived] Ratjen F, Koker P, Geller DE, Langellier-Cocteaux B, Le Maulf F, Kattenbeck S, Moroni-Zentgraf P, Elborn JS; Tiotropium Cystic Fibrosis Study Group. Tiotropium Respimat in cystic fibrosis: Phase 3 and Pooled phase 2/3 randomized trials. J Cyst Fibros. 2015 Sep;14(5):608-14. doi: 10.1016/j.jcf.2015.03.004. Epub 2015 Mar 26. PMID 25819269
- [Derived] Bradley JM, Koker P, Deng Q, Moroni-Zentgraf P, Ratjen F, Geller DE, Elborn JS; Tiotropium Cystic Fibrosis Study Group. Testing two different doses of tiotropium Respimat(R) in cystic fibrosis: phase 2 randomized trial results. PLoS One. 2014 Sep 4;9(9):e106195. doi: 10.1371/journal.pone.0106195. eCollection 2014. PMID 25188297

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomised to receive matching placebo
- Tiotropium Respimat 2.5 Micrograms: Patients randomised to receive Tiotropium Respimat 2.5 micrograms once daily
- Tiotropium Respimat 5 Micrograms: Patients randomised to receive Tiotropium Respimat 5.0 micrograms once daily
Period: Overall Study
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Started | 168 | 166 | 176
Completed | 161 | 159 | 169
Not Completed | 7 | 7 | 7
Not completed — Adverse Event | 6 | 5 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Reason discontinued not explained above | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms | Total
Number analyzed (Participants) | 168 | 166 | 176 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.4 (11.6) | 21.5 (12.0) | 20.7 (11.3) | 20.9 (11.6)
Age, Customized [Number; unit: years]
  <= 11 years | 44 | 42 | 52 | 138
  >= 12 years | 124 | 124 | 124 | 372
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 81 | 82 | 235
  Male | 96 | 85 | 94 | 275
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 2 | 3
  Black/African American | 0 | 3 | 2 | 5
  White | 127 | 124 | 132 | 383
  Missing | 39 | 35 | 37 | 111
  American Indian / Alaskan native | 2 | 3 | 3 | 8
Height [Mean (Standard Deviation); unit: centimeters] | 157.4 (17.2) | 157.7 (17.0) | 155.7 (18.2) | 156.9 (17.5)
Weight [Mean (Standard Deviation); unit: kilograms] | 52.1 (19.0) | 51.0 (17.3) | 50.4 (18.2) | 51.2 (18.1)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/square meter] | 20.3 (4.4) | 19.9 (4.0) | 20.0 (4.1) | 20.1 (4.2)
Alcohol history [Number; unit: Participants]
  Drinks no alcohol | 130 | 112 | 132 | 374
  Drinks alcohol but should not interfere with trial | 38 | 54 | 43 | 135
  Drinks alcohol but could interfere with trial | 0 | 0 | 1 | 1
Smoking history [Number; unit: Participants]
  Never smoked | 159 | 157 | 167 | 483
  Ex-smoker | 7 | 5 | 7 | 19
  Currently smokes | 2 | 4 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Predicted FEV1 AUC0-4 Response at the End of Week 12
Description: Outcome measure description: Change from baseline in percent predicted Forced Expiratory Volume in one second (FEV1) Area Under the Curve from 0 to 4 hours (AUC0-4). Calculated as percent predicted at week 12 minus percent predicted at baseline.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 163 | 158 | 169
Percentage change | -1.74 (0.65) | 1.20 (0.66) | 1.65 (0.63)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Respimat 2.5 Micrograms; Comparison of Tiotropium 2.5 microgram dose versus placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — Comment for p-value: Hierarchical testing was applied. Comparison of 2.5 dose to be performed only if superiority of tiotropium 5.0 dose compared to placebo was shown for both primary endpoints; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 2.94, 95% CI [1.19 to 4.70]
Statistical Analysis 2: Comparison: Placebo vs Tiotropium Respimat 5 Micrograms; Comparison of Tiotropium 5.0 microgram dose versus placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 3.39, 95% CI [1.67 to 5.12]

2. Primary Outcome: Percent Predicted FEV1 Trough Response at the End of Week 12
Description: Outcome measure description: Change from baseline in percent predicted trough Forced Expiratory Volume in one second. Calculated as percent predicted at week 12 minus percent predicted at baseline.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 163 | 158 | 169
Percentage change | -1.44 (0.71) | 0.81 (0.71) | 0.78 (0.69)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Respimat 2.5 Micrograms; Comparison of Tiotropium 2.5 microgram dose versus placebo; Test type: Superiority or Other; p = 0.0184, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 2.24, 95% CI [0.38 to 4.11]
Statistical Analysis 2: Comparison: Placebo vs Tiotropium Respimat 5 Micrograms; Comparison of Tiotropium 5.0 microgram dose versus placebo; Test type: Superiority or Other; p = 0.0179, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 2.22, 95% CI [0.38 to 4.06]

3. Secondary Outcome: Percent Predicted FVC AUC0-4 Response at the End of Week 12
Description: Change from baseline in percent predicted Forced Vital Capacity (FVC) Area Under the Curve from 0 to 4 hours (AUC0-4). Calculated as percent predicted at week 12 minus percent predicted at baseline.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 149 | 150 | 158
Percentage change | -1.30 (0.74) | 0.53 (0.74) | 1.81 (0.72)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Respimat 2.5 Micrograms; Comparison of Tiotropium 2.5 microgram dose versus placebo; Test type: Superiority or Other; p = 0.0756, Mixed Models Analysis; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 1.83, 95% CI [-0.19 to 3.86]
Statistical Analysis 2: Comparison: Placebo vs Tiotropium Respimat 5 Micrograms; Comparison of Tiotropium 5.0 microgram dose versus placebo; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 3.12, 95% CI [1.12 to 5.12]

4. Secondary Outcome: Percent Predicted FVC Trough Response at the End of Week 12
Description: Change from baseline in percent predicted trough Forced Vital Capacity (FVC). Calculated as percent predicted at week 12 minus percent predicted at baseline.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 149 | 150 | 158
Percentage change | -0.39 (0.73) | 0.47 (0.72) | 0.81 (0.70)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Respimat 2.5 Micrograms; Comparison of Tiotropium 2.5 microgram dose versus placebo; Test type: Superiority or Other; p = 0.3857, Mixed Models Analysis; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 0.85, 95% CI [-1.08 to 2.79]
Statistical Analysis 2: Comparison: Placebo vs Tiotropium Respimat 5 Micrograms; Comparison of Tiotropium 5.0 microgram dose versus placebo; Test type: Superiority or Other; p = 0.2199, Mixed Models Analysis; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 1.19, 95% CI [-0.72 to 3.11]

5. Secondary Outcome: Pre-bronchodilator FEF25-75 Percent Predicted at the End of Week 12
Description: Forced Expiratory Flow at 25-75% of vital capacity (FEF25-75). Calculated as percent predicted at week 12 minus percent predicted at baseline.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 150 | 152 | 158
Percentage change | -1.40 (1.57) | 2.78 (1.55) | 3.94 (1.52)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Respimat 2.5 Micrograms; Comparison of Tiotropium 2.5 microgram dose versus placebo; Test type: Superiority or Other; p = 0.0363, Mixed Models Analysis; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 4.19, 95% CI [0.27 to 8.11]
Statistical Analysis 2: Comparison: Placebo vs Tiotropium Respimat 5 Micrograms; Comparison of Tiotropium 5.0 microgram dose versus placebo; Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 5.34, 95% CI [1.45 to 9.23]

6. Secondary Outcome: Change From Baseline in Residual Volume/Total Lung Capacity (RV/TLC) at the End of Week 12
Description: Change from baseline in static lung hyperinflation as measured by RV/TLC. Calculated as percent predicted at week 12 minus percent predicted at baseline.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 53 | 54 | 54
Percentage change | -0.01 (0.03) | 0.00 (0.03) | 0.04 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Respimat 2.5 Micrograms; Comparison of Tiotropium 2.5 microgram dose versus placebo; Test type: Superiority or Other; p = 0.7414, Mixed Models Analysis; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 0.01, 95% CI [-0.06 to 0.08]
Statistical Analysis 2: Comparison: Placebo vs Tiotropium Respimat 5 Micrograms; Comparison of Tiotropium 5.0 microgram dose versus placebo; Test type: Superiority or Other; p = 0.1418, Mixed Models Analysis; Adjusted for baseline, center, visit and age group; Mean Difference (Final Values) = 0.05, 95% CI [-0.02 to 0.12]

7. Secondary Outcome: Respiratory and Systemic Symptoms Questionnaire (RSSQ)
Description: Outcome measure description: The RSSQ questionnaire is used to determine the presence or absence of an exacerbation during the recall period.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 167 | 166 | 175
Participants
  At least one pulmonary exacerbation | 16 | 13 | 12
  No pulmonary exacerbation | 151 | 153 | 163
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Respimat 2.5 Micrograms; Comparison of Tiotropium 2.5 microgram dose versus placebo; Test type: Superiority or Other; p = 0.8515, Regression, Logistic; Covariates of treatment and age group; Odds Ratio (OR) = 0.79, 95% CI [0.37 to 1.72]
Statistical Analysis 2: Comparison: Placebo vs Tiotropium Respimat 5 Micrograms; Comparison of Tiotropium 5.0 microgram dose versus placebo; Test type: Superiority or Other; p = 0.5565, Regression, Logistic; Adjusted for baseline, center, visit and age group; Odds Ratio (OR) = 0.72, 95% CI [0.33 to 1.59]

8. Secondary Outcome: Change From Baseline in CFQ Scores - Adult Group
Description: The Cystic Fibrosis questionnaire (CFQ) is a disease-specific instrument that measures health-related quality of life (HRQOL) for adults with CF. This validation questionnaire consists of 50 items on generic and disease-specific scales. The scores range from 0 to 100, with higher scores indicating better health.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 168 | 166 | 176
units on a scale
  Physical (N=99, 102, 105) | -2.5 (14.8) | -0.0 (14.1) | -2.9 (11.4)
  Role (N=94, 100, 103) | 0.7 (12.0) | -2.7 (12.0) | -2.1 (15.1)
  Vitality (N=99, 101, 105) | -2.3 (15.0) | -1.8 (16.4) | -3.3 (17.7)
  Emotion (N=99, 101, 105) | -1.1 (11.5) | -1.3 (13.5) | 0.1 (12.1)
  Social (N=99, 101, 106) | -1.1 (12.3) | -1.0 (10.7) | -0.8 (11.1)
  Body (N=99,101, 106) | 0.4 (18.4) | -0.9 (15.3) | 1.7 (16.4)
  Eat (N=99,101,106) | 1.5 (9.5) | 0.2 (10.3) | 0.0 (16.4)
  Treat (N=99, 101, 106) | 0.9 (15.5) | -1.4 (14.1) | -1.7 (12.7)
  Health (N=99, 101, 106) | -1.9 (15.1) | -3.2 (18.3) | -0.6 (18.1)
  Weight (N=95, 101, 103) | 1.4 (22.2) | -3.3 (28.9) | -0.0 (26.0)
  Respirat (N=93, 101, 103) | -1.3 (14.8) | -3.7 (15.8) | -1.8 (14.3)
  Digest (N=93, 101, 103) | 0.8 (14.9) | -1.3 (13.7) | 0.3 (14.9)

9. Secondary Outcome: Change From Baseline in CFQ Scores - Adolescents Group
Description: The Cystic Fibrosis questionnaire (CFQ) is a disease-specific instrument that measures health-related quality of life (HRQOL) for adolescents (age 6-13) with CF. This validation questionnaire consists of 50 items on generic and disease-specific scales. The scores range from 0 to 100, with higher scores indicating better health.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 168 | 166 | 176
units on a scale
  Physical (N=46, 42, 54) | 1.1 (18.0) | 3.2 (14.8) | -1.9 (15.0)
  School (N=46, 42, 55) | 1.1 (14.3) | -1.6 (10.9) | -1.1 (13.5)
  Body (N=46, 42, 55) | 2.8 (13.9) | -0.3 (16.1) | -0.1 (15.7)
  School (N=46, 42, 55) | 1.2 (18.8) | 4.2 (19.2) | 2.4 (20.9)
  Eat (N=46, 42, 55) | -1.4 (19.7) | -2.4 (17.3) | 1.6 (22.8)
  Treat (N=46, 42, 55) | 0.2 (16.5) | -1.9 (20.1) | 5.7 (19.5)
  Respirat (N=46, 42, 55) | -1.4 (15.2) | 1.2 (16.7) | -3.0 (20.2)
  Digest (N=46, 42, 55) | -5.1 (26.3) | 2.4 (26.9) | -3.0 (35.3)

10. Secondary Outcome: Change From Baseline in CFQ Scores - Parent Questionnaire
Description: The Cystic Fibrosis questionnaire (CFQ) is a disease-specific instrument that measures health-related quality of life (HRQOL) for adolescents with CF - parent questionnaire. This validation questionnaire consists of 50 items on generic and disease-specific scales. The scores range from 0 to 100, with higher scores indicating better health.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 168 | 166 | 176
units on a scale
  Physical (N=46, 45, 53) | -0.1 (15.4) | 4.9 (15.9) | 0.2 (12.7)
  Emotion (N=46, 45, 52) | -0.3 (11.2) | 0.0 (16.0) | -0.1 (15.7)
  Vitality (N=46, 44, 53) | -0.1 (12.3) | 3.3 (13.1) | -1.5 (14.9)
  School (N=46, 45, 52) | -4.8 (19.5) | 2.2 (26.3) | 0.4 (17.0)
  Eat (N=46, 43, 49) | -2.2 (23.7) | -0.8 (21.2) | 3.4 (15.9)
  Body (N=46, 45, 52) | -3.9 (18.6) | -1.7 (21.7) | -3.2 (22.6)
  Treat (N=46, 45, 52) | -2.4 (18.6) | 2.5 (16.4) | -0.2 (21.4)
  Health (N=46, 45, 52) | -2.7 (21.4) | 3.5 (23.1) | -3.0 (20.7)
  Respirat (N=45, 43, 50) | -2.8 (16.4) | -2.2 (18.8) | -6.0 (14.2)
  Digest (N=46, 43, 50) | -0.7 (15.6) | -1.8 (17.0) | 1.1 (16.8)
  Weight (N=45, 45, 49) | -5.2 (35.5) | 1.5 (30.1) | 4.1 (31.6)

11. Secondary Outcome: Amount of Tiotropium Eliminated in Urine From 0 to 4 Hours at Steady State (Ae0-4,ss)
Description: Ae0-4,ss represents the amount of tiotropium that is eliminated in urine from time 0 to 4 hours at steady state
Time Frame: pre-dose, and 5 minutes (min), 20 min, 1 hour (h), and 2 h post-dose
Population: Full Analysis Set (FAS) includes all participants having a baseline measurement and at least one post-dose measurement - patients >= 12 years
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 102 | 99
ng | 114 (73.0) | 245 (67.5)

12. Secondary Outcome: Maximum Measured Concentration at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum measured concentration of tiotropium in plasma at steady state.
Time Frame: pre-dose, and 5 minutes (min), 20 min, 1 hour (h), and 2 h post-dose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 49 | 59
pg/mL | 6.49 (58.5) | 9.95 (66.6)

13. Secondary Outcome: Time From Dosing to the Maximum Concentration (Tmax,ss)
Description: Tmax,ss represents the time from dosing to the maximum concentration of tiotropium in plasma
Time Frame: pre-dose, and 5 minutes (min), 20 min, 1 hour (h), and 2 h post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: h
Arm/Group | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 49 | 59
h | 0.0830 [0.0330 to 0.433] | 0.0830 [0.0330 to 0.333]

14. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs and Laboratory Evaluation
Description: Clinical Relevant Abnormalities for Vital Signs and Laboratory evaluation. Any new or clinically relevant worsening of baseline conditions was reported as Adverse Event.
Time Frame: From first drug administration until 30 days after last drug administration (up to 121 days)
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Number analyzed (Participants) | 168 | 166 | 176
participants
  Blood chloride decreased | 0 | 0 | 1
  Blood glucose increased | 1 | 1 | 0
  Blood pressure increased | 2 | 1 | 0
  Blood sodium decreased | 0 | 0 | 1
  Eosinophil count increased | 0 | 1 | 0
  Hepatic enzyme increased | 2 | 0 | 0
  Oxygen saturation decreased | 0 | 0 | 1
  Vitamin K decreased | 1 | 0 | 0
  White blood cell count increased | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Tiotropium Respimat 2.5 Micrograms | Tiotropium Respimat 5 Micrograms
Serious Adverse Events (participants affected / at risk) | 21/168 | 28/166 | 21/176
Other Adverse Events (participants affected / at risk) | 87/168 | 95/166 | 110/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=168) | Tiotropium Respimat 2.5 Micrograms (N=166) | Tiotropium Respimat 5 Micrograms (N=176)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cystic fibrosis (Congenital, familial and genetic disorders) | 5 | 8 | 8
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 7 | 4 | 4
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Application site hypersensitivity (General disorders) | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Overgrowth bacterial (Infections and infestations) | 1 | 0 | 0
Pleurisy viral (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Antibiotic prophylaxis (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=168) | Tiotropium Respimat 2.5 Micrograms (N=166) | Tiotropium Respimat 5 Micrograms (N=176)
Cystic fibrosis (Congenital, familial and genetic disorders) | 12 | 15 | 17
Abdominal pain (Gastrointestinal disorders) | 10 | 13 | 9
Pyrexia (General disorders) | 17 | 9 | 18
Bronchitis (Infections and infestations) | 7 | 4 | 10
Nasopharyngitis (Infections and infestations) | 14 | 11 | 14
Sinusitis (Infections and infestations) | 6 | 3 | 9
Upper respiratory tract infection (Infections and infestations) | 6 | 8 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 5 | 4
Headache (Nervous system disorders) | 18 | 7 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 34 | 46
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 5 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 9
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.